CLINICAL TRIAL: NCT00464191
Title: Escitalopram in Bipolar Depression: a Placebo-controlled Study of Acute and Maintenance Treatment
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study has been terminated because too few patients have been recruited
Sponsor: Nordfjord Psychiatric Centre (Other)
Collaborators: H. Lundbeck A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EudraCT 2005-004357-94; Lundbeck 10968; NPS 2005-1
Record Dates: First submitted 2007-04-20; First posted 2007-04-23 (Estimated); Last update posted 2009-09-21 (Estimated); Status verified 2009-09

CONDITIONS: Bipolar Disorder
Keywords: bipolar depression; SSRI; escitalopram; bipolar disorder; antidepressant; treatment trial; RCT
MeSH Terms: conditions — Bipolar Disorder | interventions — Escitalopram

INTERVENTIONS:
Drug: escitalopram

SUMMARY:
Funding: An investigator-initiated trial funded by H. Lundbeck AS.

Study design: Prospective, randomised, placebo-controlled parallel-group multicenter study.

Aim: To investigate efficacy and side effects (especially mood switches) of escitalopram,a selective serotonin reuptake inhibitor, in the acute and maintenance treatment of bipolar depression.

Hypotheses:

1. Escitalopram, given in addition to mood stabilising medications, is significantly more efficacious, measured by response and remission rates than placebo in bipolar depression (the acute phase study).
2. Continuation therapy with escitalopram gives significantly longer mean time to depressive relapse and fewer depressive relapses compared to placebo (the continuation study).
3. The incidence of "mood switching" (defined as development of mixed episodes, mania, or hypomania according to DSM-IV criteria) do not differ significantly between escitalopram and placebo in either the acute or the continuation phases.

Patients: In- and outpatients receiving care in the specialised psychiatric services of Western Norway. The population is intended to be representative of the patients treated for bipolar depression in ordinary specialist care. Patients must have a MADRS score of at least 20 at baseline. Patients with ongoing substance abuse or dependence, organic mental illness, and non-affective psychotic symptoms are excluded.

Medication: Escitalopram 10-20 mg daily or placebo in addition to mood stabilisers. The dose of mood stabilisers must have been constant for the last six weeks prior to randomisation.

Method: Phase 1 is a eight-week acute treatment trial with six clinical assessments. Patients treated with escitalopram who have not responded after eight weeks (defined by at least 50% reduction of MADRS score compared to baseline) leave the study. Placebo non-responders are treated openly with escitalopram and repeat phase 1. Responders are re-randomised to 32 weeks of maintenance treatment (phase 2). Phase 2 has nine clinical assessments. Patients who develop hypomania, mania or depressive episodes (defined as episodes meeting DSM-IV criteria for Major Depressive Episode with MADRS scores of at least 20 points) leave the study in this phase. Patients leaving the study prematurely will be offered alternative treatment.

DETAILED DESCRIPTION:
Aims

The study has two main aims:

1. To compare the efficacy and the risk of "mood switching" of escitalopram and placebo in the acute phase treatment of bipolar depression in patients already taking mood stabilising medication.
2. To compare the efficacy of escitalopram and placebo in continuation phase therapy for bipolar depression using a placebo-controlled discontinuation design. The study will compare the occurrence of syndromal and subsyndromal relapses, mixed states, mania, hypomania, and "rapid cycling" in a seven months' maintenance study following response to acute phase treatment.

Hypotheses

1. Escitalopram, given in addition to mood stabilising medications, is significantly more efficacious, measured by response and remission rates than placebo in bipolar depression (the acute phase study).
2. Continuation therapy with escitalopram gives significantly longer mean time to depressive relapse and fewer depressive relapses compared to placebo (the continuation study).
3. The incidence of "mood switching" (defined as development of mixed episodes, mania, or hypomania according to DSM-IV criteria do not differ significantly between escitalopram and placebo in either the acute or the continuation phases.

Design This is a multi-center RCT with parallel-group design. The study compares the efficacy of placebo and escitalopram, given as add-on to mood stabilising medications in patients with bipolar depression without non-affective psychotic symptoms according to DSM-IV, and with a baseline MADRS score of ≥ 20 points.

The study has two phases. The acute phase study lasts for eight weeks and compares the efficacy of escitalopram and placebo on depressive symptoms in bipolar depression. Response is defined as at least 50% improvement on the MADRS compared to the baseline score. Responders to escitalopram are re-randomised to escitalopram or placebo for the continuation phase while placebo responders continue taking placebo for the continuation phase. Patients on escitalopram who do not respond in the acute phase leave the study, whereas placebo non-responders are treated openly with escitalopram and repeat phase 1. Responders to this open-label treatment are then re-randomised double blind to escitalopram or placebo for the continuation study.

The continuation phase study lasts for 32 weeks. Patients who responded to placebo in the acute phase continue placebo and their usual mood stabilising medication for the remainder of the study. Those who responded to escitalopram are re-randomised to continue taking placebo or escitalopram in unchanged doses. Patients who develop new mood episodes (DSM-IV-defined major depressive episode, mania, hypomania, or mixed episodes) or MADRS score ≥ 20 points leave the study.

Method Screening includes sociodemographic variables, medical and psychiatric history, diagnosis made on the basis of clinical interview and verified by the MINI, symptom intensity measured by the MADRS,), results of medical examination and laboratory tests (ECG, height, weight, blood pressure and blood tests). Sociodemographic variables include age, gender, previous and concomitant disorders, course and treatment of mental disorders, bipolar disorder type (I or II), age of onset and history of psychotropic medication use.

Study procedure As soon as the blood samples are analysed, eligible patients can be randomised. They are rated on the MADRS, Clinical Global Impressions (CGI), Inventory of Depressive Symptoms - Self Report (IDS-SR), Medical Outcomes Study Short Form 12 (SF-12), Global Assessment of Functioning (GAF) and Sheehan Disability Inventory (SDI) at the baseline visit. Study medication is dispensed. The patients will return to further visits as shown below. Patients will receive study medication for a maximum of 40 weeks. Adverse events and concomitant medications are recorded.

Assessments

The following assessments will be carried out::

1. MADRS, GAF, IDS-RS, and CGI-I at week 1, 2, 4, 6, 8, 9, 10, 12, 16, 20, 24, 28, 34 and 40
2. SDI and QLDS at week 8 and 40
3. Diagnostic criteria for Mania and Hypomania at week 1, 2, 4, 6, 8, 9, 10, 12, 16, 20, 24, 28, 34 and 40
4. Diagnostic criteria for Major Depressive Episode at week 8, 9, 10, 12, 16, 20, 24, 28, 34 and 40

For the acute study, response and remission rates as assessed by the MADRS are the primary outcome measures. CGI-Improvement and IDS-SR are secondary outcome measures. In the continuation study, primary outcome measures include emergence of major depressive episodes and mania/hypomania, while time spent at different depressive symptom levels as assessed by the DSM-IV diagnostic criteria are secondary outcome measures.

Definitions Response: at least a 50% reduction of the baseline MADRS score at the end of phase 1 if the patient has completed at least four weeks of the study. CGI-I 1 or 2 at the end of phase 1.

Remission: MADRS score of 12 or less at the end of the acute phase if the patient has completed at least four weeks of the study.

New episode: A patient who has previously responded to treatment meets the DSM-IV criteria for Major Depressive Episode. The patient must score at least 15 points on the MADRS and have a CGI-S score of 3 or more during this episode.

Mania and hypomania: by DSM-IV criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bipolar disorder in major depressive episode according to DSM-IV
* MADRS score of at least 20 points at screening and baseline
* 18-70 years of age
* Unchanged dose of mood stabilising medication for at least six weeks prior to inclusion
* Voluntary, informed and written consent

Exclusion Criteria:

* Non-affective psychotic symptoms at screening
* Pregnancy or breast-feeding
* Fertile women without appropriate contraception (the pill, IUD, or contraceptive injection)
* Substance dependence during the last three months prior to baseline
* Mental retardation and organic brain disorders
* Suicide risk that mandates specific measures
* Novel (within three months) or unstable medical conditions
* Clinically significant abnormal results on medical examination or blood samples
* Exposure to escitalopram during the last three months
* Allergic reactions to citalopram or escitalopram
* Anorexia nervosa with body mass index below 18
* Formal psychotherapy started within six weeks of screening
* Electroconvulsive therapy (ECT) during the current episode of depression
* Patients who are unlikely to be reliable and compliant with study procedures
* Patients who are not fluent in Norwegian

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2006-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Phase 1:
response rates
remission rates
Phase 2:
emergence of major depressive episodes
emergence of mania, hypomania, and mixed states.

SECONDARY OUTCOMES:
Phase 1:
CGI-Improvement
change on the IDS-SR
Phase 2:
Time spent at different depressive symptom levels as assessed by the DSM-IV diagnostic criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Trond F. Aarre, MD, Principal Investigator — Nordfjord Psychiatric Centre
Locations (1):
- Nordfjord Psychiatric Centre, Nordfjordeid, Norway